CLINICAL TRIAL: NCT02418520
Title: The Effect of Miswak Chewing Sticks on the Oral Helicobacter Pylori Infection
Acronym: Miswak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Dr Jagan K Baskaradoss, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KSAUHS2015
Record Dates: First submitted 2015-04-09; First posted 2015-04-16 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Caries; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Intervention group would use Miswak chewing sticks along with the regular use of tooth brush and paste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Miswak chewing (Experimental): Chewing Sticks
  Interventions: Device: Miswak
- H.Pylori (No Intervention): Oral H.Pylori

INTERVENTIONS:
Device: Miswak — Oral hygiene with Miswak chewing sticks and normal tooth brush
  Arms: Miswak chewing

SUMMARY:
To elucidate the relationship of chewing miswak sticks on the H. Pylori infection in the oral cavity.The study would be conducted at the Faculty of Dentistry, Kuwait University.

Oral plaque samples would be obtained from those patients who are willing to participate. As a part of the initial screening the plaque samples would be collected and sent for screening of oral microbiota to the Microbiology Department of Faculty of Dentistry, Kuwait University. Here, the basic microbial culturing (rapid urease test) would be performed for detecting the presence of oral H.Pylori. Volunteers who are tested positive for H. Pylori infection through the rapid urease test would be invited to participate in the study.

DETAILED DESCRIPTION:
Ethical aspects The experimental protocol was approved by the Health Science Center (HSC) ethical committee of Kuwait University (VDR/ED/3331) and is registered at ClinicalTrials.gov as NCT02418520 (16/04/2015). Research was conducted according to the principles outlined in the declaration of Helsinki on human medical experimentation. Written informed consent was obtained from all participants and is presented in accordance to the consolidated standards of reporting trials (CONSORT) guidelines.

Study Design This was an experimental study with a randomized, cross-over, single blind design.

Study sample and Data collection This study was conducted among regular patients attending the Dental Center at Kuwait University, Kuwait. Patient recruitment started in February and was completed by the end of August 2019. The PICO (P = Patient population; I = Intervention of interest; C = Comparative intervention; O = Outcome) question for this study was, "for subjects under different fasting conditions (P), what is the effect of using miswak chewing sticks along with toothbrush (I) versus using only toothbrush (C) on the oral H. pylori counts (O)?". Volunteering patients were briefed on the study components and informed consent was obtained from them. Salivary and plaque samples were collected for PCR screening to detect the presence of H. pylori. The inclusion criteria were: 1) subjects with detectable levels of H. pylori in either plaque or salivary samples; 2) no evidence of periodontitis; and, 3) with at least 24 teeth. Subjects who received antibiotic therapy or proton-pump inhibitors within the past three months were excluded from the study.

Recruitment of study participants and grouping This study included 20 subjects who were on 12-hour fasting (fasting group) and 20 subjects who were not fasting (non-fasting group). Non-fasting group subjects were recruited between February and April and fasting group subjects were recruited between May and June 2018 (holy month of Ramadan). At baseline (T0), each subject was assigned numbers based on the chronological order of enrolment in the study. Both, the fasting and the non-fasting subjects were randomly subdivided into Group-1 and Group-2 (n=10 each). Randomized assignment of the subjects was carried out by a random binary outcome of a dice, even or odd numbers. The examiners were kept unaware of the participant allocation. Group-1 subjects were instructed to use both toothbrush and miswak (TB+M) for two weeks (T1) and only toothbrush (TB) for the next two weeks (T2); and, Group-2 subjects were asked to use only TB during T1 and TB+M during T2, for both the fasting and the non-fasting groups. Participants were given instructions on how to use miswak (five finger-grip, scrub technique, for 15 mins, twice daily21) and TB (modified Bass technique, for two minutes, twice daily) by a single investigator (JKB). Plaque and salivary samples were collected at T0, T1 and T2.

Questionnaire The subjects were interviewed and information were collected on their socio-demographic characteristics (age, gender, education, employment and income), presence of selected medical conditions (hypertension, diabetes and current medications), smoking status and dental characteristics (daily brushing frequency and previous dental visit).

Clinical Examination At baseline (T0), three trained and calibrated examiners performed the clinical examinations using a mouth mirror and a manual periodontal probe (CP11 Hu Friedy, Europe), with the patient in semi-supine position on the dental chair (A-dec, Newberg, OR, USA). The clinical examinations assessed the Silness & Löe plaque index (PI), the Löe & Silness gingival index (GI), the clinical attachment loss (CAL), the probing depth (PD) and the bleeding on probing (BOP) (inter/intra examiner reliability >80%). These measurements were performed on six surfaces (midlingual/palatal, distolingual/palatal, mesiolingual/palatal, distobuccal, midbuccal, and mesiobuccal) of all teeth. Number of missing teeth were recorded.

Sample collection procedure Plaque and salivary samples were collected from the subjects at T0, T1 and T2. Plaque samples were taken from gingival crevice at deepest pocket reading and removed from the clinical site using a sterile universal curette. The sampling area were isolated using salivary ejectors and gently dried by air. The tip of the curette was inserted into the depths of crevice/pocket, moved coronally while in contact with the tooth surface, to remove both sub and supragingival plaque. The samples were then immersed in 0.5 ml sterile distilled water in Eppendorf tubes (epTIPS Standard, Eppendorf AG, Hamburg, Germany). For the collection of stimulated salivary samples, subjects were requested to chew on paraffin wax and expectorated into a plastic funnel connected to a graded measuring cylinder. About 3 ml of saliva was collected from each subject. Immediately after collection, the sample tubes were placed in a container filled with crushed ice and transported to the Oral Microbiology lab for preserving at -800C.

Bacterial culture H. pylori JA1 strain was obtained from the Faculty of Medicine, KUWAIT University. The bacterial strain was grown on trypticase soy agar supplemented with defibrinated sheep blood (5%) at 37 degree Celsius in microaerophilic conditions.

DNA purification Saliva and plaque samples were brought to the laboratory on ice. After vortexing for 1 minute at 12000 × g, the supernatant was removed, and the pellets were stored at -80°C. DNA from the pellets was purified by using a DNeasy DNA purification Kit (Qiagen, Germany) according to manufacturer's instructions. Briefly, the pellets were treated with lysis buffer and proteinase-K at 56 degree Celsius for 1 h. DNA from lysed samples were applied onto a spin column and washed. Purified DNA was eluted using nuclease free water and the DNA concentrations were measured by UV spectrophotometry method using NanoDropTM 1000. Genomic DNA from H. pylori JA1 was purified by using the same method.

Quantitative real-time polymerase chain reaction (qPCR) After purifying the DNA from the samples, the quantities of H. pylori were measured by SYBR Green quantitative real-time PCR method using H. pylori species-specific primers for ureA gene: ureA-F: 5'-CGTGGCAAGCATGATCCAT-3' and ureA-R: 5'- GGGTATGCACGGTTACGAGTTT-3' 44. The qPCR reaction mixture (25 µl) contained 12.5 µl SYBR Green master mix (Power SYBR Green® Kit, Applied Biosystems), 1.0 µl each of forward and reverse primer (0.4 µM), 5.0 µl DNA template and 5.5 µl H2O. The thermal profile was as follows: an initial denaturation at 95°C for 10min, 40 cycles of 95°C for 15-30s, 55 °C for 30s and 72 °C for 30s. Fluorescent signal acquisition was set at the elongation step of each cycle. All qPCR reactions were run on ABpplied Biosystems® Fast 7500 Real-Time PCR machine. Sequence Detection Systems (SDS) (software version 2.3) was used for data analysis. Serially diluted genomic DNA from H. pylori JA1 was used the reactions for plotting the Ct values against deduced bacterial cell concentration (cells/mL) for each species and to construct standard curves using the above software. All the measurements were taken in triplicate for samples, standards and controls.

Data management and statistical analysis A reduction in the H. pylori count using either TB+M or TB under different fasting conditions was the primary outcome of interest in this study. As no a priori information on the effect of miswak on H. pylori was available, the sample size was calculated to detect a 50% difference between groups, assuming a mean 30% reduction in H. pylori counts between the groups, with a standard deviation of 15%. To obtain a power of 80% and for a risk alpha of 0.05, 17 patients per group were required, which was rounded-off to 20, to account for any potential dropouts. The difference in the microbial counts were computed between T0, T1 and T2. Mann-Whitney U-test or Kruskal-Wallis test (continuous dependent variable) and chi-square test (categorical dependent variable) were used to assess the differences in the general characteristics between the two groups. Distribution of H. pylori between the groups were explored for normality using the Kolmogorov-Smirnov and Shapiro-Wilk tests. The data was not normally distributed, so the intragroup change in H. pylori counts was evaluated with the Wilcoxon signed rank test and the intergroup comparisons were made using the Mann-Whitney U-test. Spearman's test was used to assess the correlation between the H. pylori counts (1x103cells/mL) in plaque/salivary samples and the clinical periodontal parameters at baseline. The level of significance was set to p<0.05. All statistical analyses were carried out using SPSS 26.0 (IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged > 18yrs
* Having >24 teeth
* Physically/mentally healthy

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The main outcome measure would be the change over time of the microbiologic data, specifically the H.Pylori counts within both groups. | 6 months
  The main outcome variable would be the change over time of the microbiologic data within both groups. Thus, the change in the number H.Pylori would be compared between the two groups at regular predetermined intervals.The patients would be recalled regularly and their plaque samples would be collected and sent for 16SrRNA gene sequencing. Gene sequencing has been known to provide more accurate information on the species of Helicobacter when compared to other methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuwait University, faculty of dentistry, Kuwait City, Kuwait

REFERENCES:
- [Background] Rifaey N, AlAdwani M, Karched M, Baskaradoss JK. A clinical investigation into the efficacy of miswak chewing sticks as an oral hygiene aid: A crossover randomized trial. Int J Dent Hyg. 2021 May;19(2):223-230. doi: 10.1111/idh.12484. Epub 2020 Dec 20. PMID 33258168
- [Background] Aksit Bicak D, Akyuz S, Kiratli B, Usta M, Urganci N, Alev B, Yarat A, Sahin F. The investigation of Helicobacter pylori in the dental biofilm and saliva samples of children with dyspeptic complaints. BMC Oral Health. 2017 Mar 21;17(1):67. doi: 10.1186/s12903-017-0361-x. PMID 28327128
- [Result] Contractor QQ, Tahir MY, Naseem S, Ahmad S. Helicobacter pylori in the dental plaque of healthy Saudis. Saudi J Gastroenterol. 1998 Jan;4(1):13-6. PMID 19864780